CLINICAL TRIAL: NCT04241692
Title: Comparative Study of the CarnationTM Ambulatory Monitoring Sternal ECG Patch System With a Conventional 24-Hour 7 Lead Holter Monitor Recorder
Brief Title: Comparative Study of the Sternal Patch System With a Conventional Holter Recorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Jeffrey Moak, Jeffrey P. Moak, MD, Director, Electrophysiology and Pacing; Principle Investigator, Professor of Pediatrics, Children's National Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00013642
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Cardiac Arrhythmia; Syncope
MeSH Terms: conditions — Arrhythmias, Cardiac; Syncope

STUDY DESIGN:
Intervention Model Description: To allow for this type of comparison, each enrolled research subject will wear both systems simultaneously
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Application of Carnation Ambulatory Patch Monitoring System (Experimental): The patient will wear a Standard Holter Monitor and the CAM Patch system simultaneously for 24 hours.
  Interventions: Device: CarnationTM Ambulatory Monitoring Sternal ECG Patch System
- Application Conventional 24-Hour Holter Monitor Recorder (Experimental): The patient will wear a Standard Holter Monitor and the CAM Patch system simultaneously for 24 hours.
  Interventions: Device: Conventional 24-Hour 7 Lead Holter Monitor Recorder

INTERVENTIONS:
Device: CarnationTM Ambulatory Monitoring Sternal ECG Patch System — A newly developed cardiac rhythm monitoring system
  Arms: Application of Carnation Ambulatory Patch Monitoring System
Device: Conventional 24-Hour 7 Lead Holter Monitor Recorder — Traditional recordings made using a standard 24-hour Holter monitor.
  Arms: Application Conventional 24-Hour Holter Monitor Recorder

SUMMARY:
This study will be a comparison of two externally worn recording systems for documentation of cardiac arrhythmias in symptomatic patients or patients at risk for arrhythmia. Non-invasive documentation of cardiac arrhythmias can be done using the standard electrocardiogram (ECG). This has limitations given it is performed for only a 10 sec period. Alternative methods for making longer term recording have been developed. The standard device is the 24 hour 7-lead Holter monitor. Newer technology has simplified the hardware needed to make these longer term recordings, and incorporate a self-contained recording system in a patch that is applied over the patient's chest. Little is known comparing the sensitivity, specificity and recording noise / signal artifact between the older technology (standard 24-Hour Holter monitor) and the Patch electrode.

DETAILED DESCRIPTION:
Objective: Comparison of two externally worn recording systems for documentation of cardiac arrhythmias in symptomatic patients or patients at risk for arrhythmia. Non-invasive documentation of cardiac arrhythmias can be done by attempting to take a snapshot view of a patient's cardiac rhythm using the standard electrocardiogram (ECG). This has limitations given it is performed for only a 10 sec period, and requires the patient to be symptomatic at the time of the recording. Therefore, the sensitivity of this technique is very low. Alternative methods for making longer term recording have been developed and used for decades. The standard device is the 24 hour 7-lead Holter monitor. These devises are large, restrict patient mobility and require cables to be connected between the applied skin ECG electrodes placed on the patient's chest and the recording device. Newer technology has simplified the hardware needed to make these longer term recordings, and incorporate a self-contained recording system in a patch that is applied over the patient's chest. These units allow for unlimited mobility, are significantly smaller, easier to wear and have eliminated the requirement for cables to connect the electrodes with the recording device. However, little is known comparing the sensitivity, specificity and recording noise / signal artifact between the older technology (standard 24-Hour Holter monitor) and the Patch electrode.

Specific Aims:

Aim 1: Comparison of Cardiac Arrhythmia Documentation between Standard 24-Hour Holter Monitor vs. Patch Monitor To evaluate the diagnostic yield for cardiac arrhythmias between the two recording systems.

The presence and frequency (qualitative and quantitative) of cardiac arrhythmias documented by each recording system with be compared. To allow for this type of comparison, each enrolled research subject with wear both systems simultaneously.

Aim 2: Comparison of Recording Quality between Standard 24-Hour Holter Monitor vs. Patch Monitor To evaluate percentage of time ECG signal quality is poor and uninterpretable.

Aim 3: Comparison of Comfortability Between Standard 24-HourHolter Monitor vs. Patch Monitor Recording Quality To evaluate level of patient's discomfort during the application of each recording system. Since both systems will be applied at the same time it may be hard for the research subject to rank the comfortability of the two systems. We will focus in this aim at more objective measures such as skin irritation under the recording electrodes, and frequency of time during which the skin electrodes come off the patient and require re-application.

Hypotheses:

Aim 1: Comparison of Cardiac Arrhythmia Documentation between Standard 24-Hour Holter Monitor vs. Patch Monitor We hypothesize that there will be no qualitative or quantitative difference in arrhythmia frequency between the two recording techniques, i.e. that both devices will detect all spontaneous arrhythmias with similar quantitative counts of ectopic beats (+/- 5%).

Aim 2: Comparison of Recording Quality between Standard 24-Hour Holter Monitor vs. Patch Monitor We hypothesize that recording quality will be better with the Patch Monitor since there are not 7 separately applied skin electrodes and cables connecting the electrodes with the recorder, resulting in a lower percent of poor ECG signal quality.

Aim 3: Comparison of Comfortability Between Standard 24-hour Holter Monitor vs. Patch Monitor Recording Quality We hypothesize that the degree of skin irritation and level of discomfort in the region of application will be less with the Patch Monitor. We hypothesize that the ECG leads will fall off from its site of application will be less with the Patch Monitor.

ELIGIBILITY:
Inclusion Criteria:

* Any infant, child, adolescent, or young adult with one or more of the following:

  1. Syncope
  2. Pre-syncope
  3. Palpitations
  4. Management of a known or suspected cardiac arrhythmia

Exclusion Criteria:

* Any inflamed or friable skin over the anterior thorax and upper abdomen or a sternal incision within 3 months from the date of enrollment

Max Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Difference in Cardiac Arrhythmia Detection Between Recording Systems | 24 Hours
  The presence (yes/no) and frequency of cardiac arrhythmias will be quantitated on each recording system for comparison
Difference in Signal Quality Between Recording Systems | 24 Hours
  We will quantitatively evaluate percentage of time signal quality is poor and uninterpretable with each recording system.

SECONDARY OUTCOMES:
Difference in Skin Discomfort Between Recording Systems | 24 Hours
  User will rate skin discomfort on a pre-determined scale: none, mild, moderate, severe at each site of application

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bigger JT Jr, Reiffel JA, Coromilas J. Ambulatory electrocardiography. In: Platia E, ed. Non-Pharmacologic Management of Cardiac Arrhythmias. Philadelphia: JB Lippincott, 1986:36-61.
- [Background] Clark PI, Glasser SP, Spoto E Jr. Arrhythmias detected by ambulatory monitoring. Lack of correlation with symptoms of dizziness and syncope. Chest. 1980 Jun;77(6):722-5. doi: 10.1378/chest.77.6.722. PMID 7398383
- [Background] Gibson TC, Heitzman MR. Diagnostic efficacy of 24-hour electrocardiographic monitoring for syncope. Am J Cardiol. 1984 Apr 1;53(8):1013-7. doi: 10.1016/0002-9149(84)90628-3. PMID 6702676
- [Background] Heilbron EL. Advances in modern electrocardiographic equipment for long-term ambulatory monitoring. Card Electrophysiol Rev. 2002 Sep;6(3):185-9. doi: 10.1023/a:1016322218490. PMID 12114836
- [Background] Jonas S, Klein I, Dimant J. Importance of Holter monitoring in patients with periodic cerebral symptoms. Ann Neurol. 1977 May;1(5):470-4. doi: 10.1002/ana.410010511. PMID 363045
- [Background] Kapoor WN, Cha R, Peterson JR, Wieand HS, Karpf M. Prolonged electrocardiographic monitoring in patients with syncope. Importance of frequent or repetitive ventricular ectopy. Am J Med. 1987 Jan;82(1):20-8. doi: 10.1016/0002-9343(87)90372-x. PMID 2432783
- [Background] Zimetbaum P, Josephson ME. Evaluation of patients with palpitations. N Engl J Med. 1998 May 7;338(19):1369-73. doi: 10.1056/NEJM199805073381907. No abstract available. PMID 9571258